CLINICAL TRIAL: NCT06181227
Title: A Phase 2 Study to Evaluate the Safety and Treatment Effect of Intravitreal AVD-104 in Participants With Diabetic Macular Edema
Brief Title: A Phase 2 Study of Intravitreal AVD-104 in Diabetic Macular Edema
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped early due to insufficient study drug supply and study funding constraints
Sponsor: Aviceda Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVD-104-C301
Record Dates: First submitted 2023-11-28; First posted 2023-12-26 (Actual); Results first posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose AVD-104 (Experimental): Three intravitreal injections at 1.0 milligram per eye each 28 days apart will be administered to the study eye. Participants will be followed for 84 days total.
  Interventions: Drug: AVD-104
- High dose AVD-104 (Experimental): Two intravitreal injections at 2.0 milligrams per eye 56 days apart will be administered to the study eye. Participants will be followed for 84 days total.
  Interventions: Drug: AVD-104

INTERVENTIONS:
Drug: AVD-104 — An intravitreal injection of 50 microliters at the doses described will be given. Visual acuity, optical coherence tomography thickness and vascular perfusion will be evaluated for an effect of the drug.

SUMMARY:
A Phase 2 study to determine the safety and preliminary efficacy of intravitreal injections of AVD-104, a novel glyco-mimetic nanoparticle, in reducing macular edema associated with diabetic retinopathy.

DETAILED DESCRIPTION:
The primary objective is to evaluate the tolerability and treatment effect of intravitreal injections (IVT) of AVD-104 in participants with diabetic macular edema (DME). Participants will receive either three intravitreal injections of low-dose AVD-104 (1.0 mg) each 28 days apart or two intravitreal injections of AVD-104 at a high-dose (2.0 mg) 56 days apart. Serial optical coherence tomography (OCT), ultra wide-field fluorescein angiography, and OCT-angiography (OCT-A) will be performed to evaluate the treatment effect on central subfield thickness (CST) and areas of non-perfusion. All participants will be followed-up for safety until day 84.

There will be a planned enrollment up to 30 participants.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or 2), as defined by the World Health Organization and/or American Diabetes Association
* Decreased visual acuity (VA) due to DME, with Best corrected visual acuity (BCVA) letter score of 75-20 letters on ETDRS-like charts (20/32-20/320 Snellen equivalent)
* DME represented by macular thickening on Spectral domain optical coherence tomography (SD-OCT) involving the center of the macula: Central subfield thickness (CST) ≥325 μm

Exclusion Criteria:

* Any IVT anti-vascular endothelial growth factor (VEGF) treatment within 3 months before randomization
* Any history of pan-retinal photocoagulation (PRP) treatment
* Any use of Iluvien® (Alimera Sciences, Inc., Alpharetta, GA) in the last 3 years; or Ozurdex® (Abbvie, Chicago, IL) or Xipere (Bausch & Lomb, Vaughan, Ontario, Canada) in the last 6 months
* History of macular laser photocoagulation
* Any signs of high-risk proliferative diabetic retinopathy (PDR)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Callanan, MD, Study Director — Aviceda Therapeutics
Locations (3):
- United States (3):
  - Erie Retina Research, Erie, Pennsylvania
  - Texas Retina Associates, Dallas, Texas
  - West Texas Retina Consultants, Wichita Falls, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose AVD-104 | High Dose AVD-104
Started | 10 | 11
Completed | 3 | 2
Not Completed | 7 | 9
Not completed — Study terminated by sponsor | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose AVD-104 | High Dose AVD-104 | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.44) | 66.6 (11.14) | 66.0 (9.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 2 | 5 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: American Indian or Alaska Native | 1 | 0 | 1
  Ethnicity: Black or African American | 2 | 0 | 2
  Ethnicity: White | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of participants with any evidence of serious adverse events as assessed by ocular examination
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose AVD-104 | High Dose AVD-104
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

2. Secondary Outcome: Treatment Effect
Description: Evaluate the treatment effect of AVD-104 at multiple doses on central subfield thickness (CST) as measured by Spectral-domain optical coherence tomography (SD-OCT)
Time Frame: 3 months
Population: The trial was discontinued due to Intellectual property (IP) supply issues and study funding constraints. Only 6 participants received treatment with scheduled follow-up to 3 months and gradable SD-OCT. The planned treatment schedule for 30 participants was not achieved.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Low Dose AVD-104 | High Dose AVD-104
Number analyzed (Participants) | 2 | 4
microns
  Baseline | 653.5 (116.7) | 432.0 (111.8)
  Month 3 | 803.5 (10.6) | 560.3 (254.1)

3. Secondary Outcome: Treatment Effect - Vision
Description: Evaluate the treatment effect of AVD-104 at multiple doses on Best-corrected visual acuity (BCVA) using ETDRS ((Early-Treatment Diabetic Retinopathy Study) visual acuity charts
Time Frame: 3 months
Population: The trial was discontinued due to IP supply issues and study funding constraints. Only 6 participants received treatment up to 3 months of the planned 30 participants. 10 of the participants only received a single injection. This is a limited sample and the planned treatment schedule was not achieved.
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Low Dose AVD-104 | High Dose AVD-104
Number analyzed (Participants) | 2 | 4
ETDRS letters
  Baseline | 52 (11.3) | 67 (9.8)
  Month 3 | 25.5 (0.7) | 68 (16.3)

ADVERSE EVENTS:
Time Frame: The first participant was enrolled 11-30-2023 with last participant visit on 04-05-2024. The study was terminated early with only 7 participants followed for the planned 3 month followup period. 13 of the remaining participants were seen for an early close-out safety visit with 1 participant lost to followup.
Arm/Group | Low Dose AVD-104 | High Dose AVD-104
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 5/10 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose AVD-104 (N=10) | High Dose AVD-104 (N=11)
Visual impairment (Eye disorders) | 2 (2) | 0 (0)
Eye inflammation (Eye disorders) | 2 (3) | 0 (0)
Vitreous opacities (Eye disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/27/NCT06181227/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT06181227/SAP_001.pdf